CLINICAL TRIAL: NCT02113423
Title: Superiority of Intensity Modulated Radiotherapy in Recurrent T1-2 Nasopharyngeal Carcinoma
Brief Title: Intensity Modulated Radiotherapy in Recurrent T1-2 Nasopharyngeal Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FJCH009911
Record Dates: First submitted 2014-04-08; First posted 2014-04-14 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Nasopharyngeal Cancer Recurrent
Keywords: superiority, re-irradiation, IMRT, recurrent T1-2 NPC
MeSH Terms: interventions — Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- recurrent T1-2 NPC,no treatment (Experimental): 3D-CRT, IMRT, BT, BT combined 3D-CRT or IMRT
  Interventions: Radiation: 3D-CRT, IMRT, BT, BT combined 3D-CRT or IMRT

INTERVENTIONS:
Radiation: 3D-CRT, IMRT, BT, BT combined 3D-CRT or IMRT — 3D - CRT（3D-Conformal Radiotherapy）: CTV-P 50-60Gy(2 Gy or 1.8 Gy per daily fraction, 5 days per week) IMRT（Intensity Modulated Radiotherapy）: GTV-P 50-60 Gy(2 Gy or 1.8 Gy per daily fraction, 5 days per week) BT(Brachytherapy): 2.5Gy BID*10F one week interval BT combined 3D - CRT or IMRT: First,GTV-P 40Gy(2 Gy or 1.8 Gy per daily fraction, 5 days per week);Then, 2.5Gy BID*2F

SUMMARY:
The hypothesis of the study is to address the efficacy and toxicity profile of aforementioned four modalities for rT1-2 NPC.

Characters of the patients:

* list item one: 168 patients, median age 48 years (range 16-75 years） proven rT1-2 NPC were diagnosed
* list item two: Treated with four different irradiation modalities(3D-CRT,IMRT, BT , BT Combined 3D-CRT or IMRT).
* list item three: Median time to recurrence was 30 months (range 1-180months). The median follow-up time was 28 months (range, 4-135 months).

DETAILED DESCRIPTION:
Objectives:

Recurrent T1-2 Nasopharyngeal Carcinoma (rT1-2) may be salvaged by 3D - CRT（3D-Conformal Radiotherapy）, IMRT（ Intensity Modulated Radiotherapy）, Brachytherapy (BT), BT combined 3D - CRT or IMRT . The aim of this study is to address the efficacy and toxicity profile of aforementioned four modalities for rT1-2 NPC.

Methods and Materials:

168 patients, median age 48 years (range 16-75 years） proven rT1-2 NPC were diagnosed and treated with four different irradiation modalities(3D-CRT,IMRT, BT , BT Combined 3D-CRT or IMRT) . Median time to recurrence was 30 months (range 1-180months). The median follow-up time was 28 months (range, 4-135 months).

ELIGIBILITY:
Inclusion Criteria:

* recurrent T1-2 nasopharyngeal carcinoma patients

Exclusion Criteria:

* non recurrent T1-2 nasopharyngeal carcinoma patients

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 1996-01; Primary Completion 2009-06 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
all cause mortality | thirteen years

CONTACTS AND LOCATIONS:
Overall Officials: Jianji Pan, MD, Study Director — Department of Radiation Oncology, Cancer Hospital of Fujian Medical University, Fuzhou, Fujian, People's Republic of China
Locations (1):
- Fujian Cancer Hospital Radiation Oncology Department, Fuzhou, Fujian, China